CLINICAL TRIAL: NCT05719168
Title: Exploring the Role of Gastric Neuromuscular Function in the Pathophysiology of Proton Pump Inhibitor (PPI) Refractory Gastresophageal Reflux Disease (GERD)
Brief Title: Gastric Neuromuscular Function in GERD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Functional Gut Clinic (Other)
Responsible Party: Principal Investigator, Dr Anthony Hobson, Clinical Director, The Functional Gut Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: FGC-22-002
Record Dates: First submitted 2022-08-30; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: GERD
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Intervention Model Description: Prospective, cross-sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients with medical refractory GERD (Experimental): Participants undergo BSGM for 4.5 hours with simultaneous oesophageal manometry, pH-impedance monitoring and gastric emptying breath tests. Following completion, participants continue with ambulatory pH-impedance monitoring for a further 24-hours.
  Participants undergo a hydrogen and emthane breath test on a seperate day.
  Interventions: Device: Body Surface Gastric Mapping
- Healthy controls without gastrointestinal symptoms (Active Comparator): Participants undergo BSGM for 4.5 hours with simultaneous oesophageal manometry, pH-impedance monitoring and gastric emptying breath tests. Following completion, participants continue with ambulatory pH-impedance monitoring for a further 24-hours.
  Interventions: Device: Body Surface Gastric Mapping

INTERVENTIONS:
Device: Body Surface Gastric Mapping — 64-channel electrode array placed on the outer abdomen

SUMMARY:
Bodysurface gastric mapping (BSGM) will be used to assess gastric neuromuscular function in healthy controls and patients with medical refractory gastroesophageal reflux disease (GERD).

Participants will undergo BSGM for 4-hours in addition to high resolution manometry (HRM), pH-impedance monitoring, and gastric emptying breath test.

DETAILED DESCRIPTION:
This is a clinical trial of a non-invasive BSGM medical device (Gastric Alimetry) in patients with medical refractory GORD and healthy controls to determine the differences in gastric electrical activity, and correlate with adjacent measurements of gastro-esophageal function.

Patients referred to the Functional Gut Clinic for standard care investigation of GORD with HRM and pH-impedance monitoring will be recruited. Healthy volunteers will be recruited via advertisement.

All patients and healthy volunteers will undergo BSGM at the research site, which lasts around 4.5 hours. After a 0.5 hour baseline, subjects will undergo HRM and pH-impedance monitoring concomitantly. A test meal of porridge with C13 labelled octanoic acid will be consumed with BSGM and breath samples recorded for 4.0 hours after meal completion. The HRM catheter will be removed after 1.0 hour from finishing the test meal whist the pH-impedance monitoring will continue for the remainder of the site visit and for the remainder of the 24-hour study period whilst the subject is at home to quantify reflux.

ELIGIBILITY:
Healthy controls

Inclusion Criteria:

* Aged 18-70 years old
* BMI 18-35
* Able to understand written and spoken English
* Able to provide written consent
* Able to understand risks and benefits

Exclusion Criteria:

* Antacid use (e.g. PPI, H2RA or Gaviscon) within last 12-months
* Active use of other medications known to impact gastric motility
* Upper GI symptoms including but not limited to heartburn, regurgitation, epigastric pain, nausea and bloating
* Significant medical condition
* History of skin allergies or hypersensitivity
* Active abdominal wounds or abrasions, fragile skin
* Current pregnancy
* Vulnerable group e.g. prisoners/cognitive impairment/institutionalised individuals
* Regular cannabis users (unable to abstain for 7-days)
* Opioid user
* Unable to use a tablet device

GORD patients

Inclusion Criteria

* Referred for 24-hour pH-impedance monitoring
* Aged 18-70 years old
* BMI 18-35
* Able to understand written and spoken English
* Able to provide written consent
* Able to understand risks and benefits

Exclusion Criteria

* Systemic or metabolic disorder known to cause gastric dysmotility other than diabetes (e.g. scleroderma, multiple sclerosis, hyperthyroidism).
* History of upper GI surgery or hiatal hernia (>5cm, paraesophageal, or 'large' on endoscopy report)
* Diabetic and on insulin
* Proven mechanical bowel obstruction
* History of skin allergies or hypersensitivity
* Active abdominal wounds or abrasions, fragile skin
* Current pregnancy
* Vulnerable group - prisoners/cognitive impairment/institutionalised individuals
* Regular cannabis users (unable to abstain for 7-days)
* Opioid user
* Unable to use a tablet device

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Difference in BSGM parameters between GORD and healthy controls | 24-hours
  Gastric Alimetry Rhythm Index (Normal >0.25)
Difference in BSGM parameters between GORD and healthy controls | 24-hours
  Prinicpal Gastric Frequency (Normal: 2.65-3.35cpm)
Difference in BSGM parameters between GORD and healthy controls | 24-hours
  Fed:Fasted Amplitude ratio (Normal: >1.08)
Difference in BSGM parameters between GORD and healthy controls | 24-hours
  Average Amplitude (Normal: 20-70 microvolts)
Difference in BSGM parameters between GORD and healthy controls | 24-hours
  % of retrograde activity

SECONDARY OUTCOMES:
Normal reference ranges for gastric emptying and BSGM | 24-hours
  T lag and T 1/2 time (minutes)
Correlate reflux event frequency with Gastric Alimetry Rhythm Index | 24-hours
  Frequency of reflux events with Gastric Alimetry Rhythm Index
Correlate reflux event frequency with Prinicpal Gastric Frequency (cpm) | 24-hours
  Frequency of reflux events with Prinicpal Gastric Frequency (cpm)
Correlate reflux event frequency with Fed:Fasted Amplitude ratio | 24-hours
  Frequency of reflux events with Fed:Fasted Amplitude ratio
Correlate reflux event frequency with Average Amplitude | 24-hours
  Frequency of reflux events with Average Amplitude (microvolts)
Correlate reflux event frequency with % of retrograde activity | 24-hours
  Frequency of reflux events with % of retrograde activity
Correlate symptom severity with BSGM parameters | 24-hours
  Real time discrete (vomiting, belching, reflux counts) and continuous (Nausea, bloating, upper gut pain, heartburn, stomach burn and excessive fullness) gastrointestinal symptom scores at both pre- and post-prandial time periods determined by a series of multiple 10-point symptom severity scales integrated within the validated Gastric Alimetry iOS Application with Gastric Alimetry Rhythm Index
Correlate quality of life with BSGM parameters | 24-hours
  Total symptom burden scores according to the PAGI-QOL with Gastric Alimetry Rhythm Index
Correlate the results of gastric emptying with BSGM parameters | 24-hours
  T lag and T 1/2 (minutes) with ith Gastric Alimetry Rhythm Index
Correlate the results of oesophageal manometry with BSGM parameters | 24-hours
  Distal contractile integral (mmHg.s.cm) with Gastric Alimetry Rhythm Index
Correlate the results of oesophageal manometry with Gastric Alimetry Rhythm Index | 24-hours
  Integrated relaxation pressure (mmHg) with Gastric Alimetry Rhythm Index
Correlate the results of oesophageal manometry with Prinicpal Gastric Frequency | 24-hours
  Integrated relaxation pressure (mmHg) with Prinicpal Gastric Frequency
Correlate the results of oesophageal manometry with Prinicpal Gastric Frequency | 24-hours
  Integrated relaxation pressure (mmHg) with % of retrograde activity
Correlate the results of oesophageal manometry with Gastric Alimetry Rhythm Index | 24-hours
  Frequency of transient lower oesophageal sphincter relaxation (TLOSRs) with Gastric Alimetry Rhythm Index
Correlate the results of oesophageal manometry with Gastric Alimetry Rhythm Index | 24-hours
  Frequency of transient lower oesophageal sphincter relaxation (TLOSRs) with Prinicpal Gastric Frequency
Correlate the results of oesophageal manometry with % of retrograde activity | 24-hours
  Frequency of transient lower oesophageal sphincter relaxation (TLOSRs) with % of retrograde activity
Correlate the results of hydrogen and methane breath testing with Gastric Alimetry Rhythm Index | 7 days
  Total gas production (AUC ppm) with Gastric Alimetry Rhythm Index

CONTACTS AND LOCATIONS:
Locations (1):
- The Functional Gut Clinic, Manchester, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No